CLINICAL TRIAL: NCT06714305
Title: Comparison of Effectiveness of Hand Versus Rotary Instrumentation in Pulpectomy of Primary Second Molar Teeth.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RANA AHMAD (Other)
Responsible Party: Sponsor-Investigator, RANA AHMAD, Investigator, Assistant professor (Clinical), Depatment of Operative dentistry, School of dentistry, Shaheed Zulfiqar Ali Bhutto Medical University
Organization: Shaheed Zulfiqar Ali Bhutto Medical University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CPSP/REU/2014-077-1257
Record Dates: First submitted 2024-11-22; First posted 2024-12-03 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Irreversible Pulpitis (toothache)
MeSH Terms: conditions — Toothache

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Group A will be assigned to hand instrumentation. (Active Comparator): the canal will be prepared by hand hedstorm files, manually by step back technique.
  Interventions: Device: will be assigned to rotary instrumentation.
- rotary instrumentation of primary second molar tooth (Experimental): NiTi rotary protaper system will be used for canal preparation by crown down technique in primary second molar tooth
  Interventions: Device: Group B will be assigned to rotary instrumentation.

INTERVENTIONS:
Device: Group B will be assigned to rotary instrumentation. — group B, NiTi rotary protaper system will be used for canal preparation by crown down technique.
  Arms: rotary instrumentation of primary second molar tooth
Device: will be assigned to rotary instrumentation. — the canal will be prepared by conventional hedstorm files manually by step back technique.
  Arms: Group A will be assigned to hand instrumentation.

SUMMARY:
To provide an effective technique for pulpectomy in primary second molar teeth in pakistani population, local studies are required. No local studies have been done so far and limited number of international in vivo studies have been conducted previously. Hence this study will evaluate the effectiveness of this technique in pakistani population. If results of this study will be significant in favor of this technique, it will be applied with confidence in same population. There will be better compliance of patients as procedure will be done in single visit.

ELIGIBILITY:
Inclusion Criteria:

1. Children of both genders having age 4-6.5 years
2. Children having signs and symptoms of irreversible pulpitis in their second primary molar teeth on clinical examination as per operational definition.

Exclusion Criteria:

1. Children having previously accessed pulpectomy assessed clinically and on periapical radiographs.
2. Children having acute/chronic abcesses in teeth under consideration seen clinically.
3. Children having furcal or periapical radiolucency around teeth under consideration seen on periapical radiograph.
4. Diabetic, haemophilic or medically compromised children found on history
5. Children who fail to attend appointments.

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
To compare the effectiveness of manual versus rotary instrumentation for pulpectomy in primary second molar teeth irreversible pulpitis | immediately after obturation
  Effectiveness of instruments will be determined by analyzing the adequacy of root canal filling. Adequacy will be checked immediately after root canal filling on periapical radiographs by measuring with scale the distance of root canal filling from apex to length of filling material in both mesial and distal roots. If distance is less than 2.5 mm, it will be called as effective.

CONTACTS AND LOCATIONS:
Locations (1):
- Nishter Institute of Dentistry, Multan, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided